CLINICAL TRIAL: NCT01477333
Title: An Evaluation of the Safety and Efficacy of the Addition of UT-15C SR to Pulmonary Arterial Hypertension Patients Currently Receiving Tyvaso®
Brief Title: Addition of UT-15C SR to Pulmonary Arterial Hypertension Patients Currently Receiving Tyvaso®
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDE-PH-203
Record Dates: First submitted 2011-11-14; First posted 2011-11-22 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2017-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Tyvaso; UT-15C SR; PAH
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UT-15C SR BID (Experimental): Initiated at 0.125 mg twice daily (BID), titrated as clinically indicated.
  Interventions: Drug: UT-15C SR; Drug: Tyvaso Inhalation Solution

INTERVENTIONS:
Drug: UT-15C SR — Initiated at 0.125 mg BID, titrated as clinically indicated.
  Other Names: treprostinil diethanolamine, sustained release
Drug: Tyvaso Inhalation Solution — Administered as at least 9 breaths 4 times daily for at least 4 weeks prior to Baseline
  Other Names: Treprostinil

SUMMARY:
The purpose of this multi-center, open-label, safety and tolerability study was to assess the addition of oral treprostinil (UT-15C sustained release [SR] tablets) to subjects currently receiving Tyvaso (treprostinil) inhalation solution. During the 24-week evaluation period, the study evaluated the changes in the following assessments: hemodynamics, 6-minute walk test (6MWT), Borg dyspnea score, N-Terminal pro-brain natriuretic peptide (NT-proBNP), World Health Organization (WHO) Functional Class, and safety assessments.

Eligible subjects had a diagnosis of pulmonary arterial hypertension (PAH), currently were receiving Tyvaso, and may have been receiving other approved PAH specific oral therapies (endothelin receptor antagonists [ERAs] and/or phosphodiesterase type 5 inhibitor [PDE5-I], if at a stable dose for ≥30 days). At Baseline, subjects received the first dose of 0.125 mg UT-15C SR.

DETAILED DESCRIPTION:
This was a multi-center, open-label, safety and tolerability study in WHO Group 1 PAH subjects adding UT-15C SR to Tyvaso and PAH approved background therapy. This study had a 24-week evaluation period followed by a long term safety period. Six study visits occurred in the first 24 weeks of study; Screening, Baseline, Week 4, Week 8, Week 12, and Week 24 visits. Right heart catheterization occurred between 2-4 hours following the last Tyvaso dose at Baseline (prior to the administration of UT-15C SR) and Week 24.

ELIGIBILITY:
Significant inclusion criteria included:

1. Subjects were between 18 to 75 years of age
2. Diagnosis of PAH: Idiopathic; Heritable; Associated with: Collagen vascular disease, Human immunodeficiency virus (HIV) infection, appetite suppressant or toxin use, or repaired congenital systemic-to-pulmonary shunts (repaired ≥5 years)
3. Had been receiving Tyvaso for at least 4 weeks (≥9 breaths, 4 times a day [QID]) and required additional therapy
4. In addition to Tyvaso, subjects may have been receiving other approved PAH specific oral therapies (ERAs and/or PDE-5 inhibitors, if at a stable dose)

Significant exclusion criteria included:

1. The subject was pregnant or lactating
2. The subject had previously received UT-15C SR
3. The subject had added, discontinued or changed the dosing regimen (i.e., prescription) of conventional PAH therapies (e.g., oral vasodilators, oxygen, digoxin) within 21 days of Baseline
4. The subject was receiving a FDA approved PAH therapy (e.g., ERA and/or PDE-5 inhibitor) for less than 30 days prior to Baseline, or the dose had been modified within 30 days of Baseline
5. The subject had any disease associated with PAH other than collagen vascular disease, HIV infection, repaired congenital systemic-to-pulmonary shunts (for at least 5 years), or appetite suppressant/toxin use (e.g., portal hypertension, chronic thromboembolic disease, pulmonary veno-occlusive disease, etc.), or had an atrial septostomy
6. The subject had ischemic heart disease prior to Screening, or left ventricular dysfunction as evidenced by a mean PCWP (or a left ventricular end diastolic pressure) greater than 15 mmHg or left ventricular ejection fraction (LVEF) less than 40% as assessed by either multigated angiogram (MUGA), angiography or echocardiography. Patients with abnormal left ventricular function attributable entirely to impaired left ventricular filling due to the effects of right ventricular overload were not excluded.
7. The subject had uncontrolled systemic hypertension as evidenced by systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than 100 mmHg at Baseline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Madden, MD, MPH, Study Chair — Associate Director, Medical Development
Locations (6):
- United States (6):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this study was October 2011 to November 2013.
Period: Overall Study
Arm/Group | UT-15C SR BID
Started | 18
Completed | 15
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Clinical Deterioration | 1

BASELINE CHARACTERISTICS:
Arm/Group | UT-15C SR BID
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 51.3 [20 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemodynamic Parameters From Baseline to Week 24.
Description: Hemodynamics (via right heart catheterization [RHC]) were assessed at Baseline and Week 24 or at the time of premature termination of study drug if prior to the Week 24 visit.
  Cardiopulmonary hemodynamic measurements included the following: mean pulmonary arterial pressure (PAPm), mean systemic arterial pressure (SAPm), mean right atrial pressure (RAPm), and mean pulmonary capillary wedge pressure (PCWPm).
Time Frame: Baseline and Week 24
Population: Intent-to-treat population with data available at Baseline and Week 24.
Measure: Median (Full Range); unit: mmHg
Arm/Group | UT-15C SR BID
Number analyzed (Participants) | 15
mmHg
  Systolic systemic arterial pressure (mmHg) | -2.0 [-22 to 21]
  Diastolic systemic arterial pressure (mmHg) | 0 [-20 to 18]
  Mean systemic arterial pressure (mmHg) | -1.0 [-29 to 18]
  Systolic pulmonary arterial pressure (mmHg) | 3.0 [-51 to 12]
  Diastolic pulmonary arterial pressure (mmHg) | 0 [-16 to 10]
  Mean pulmonary arterial pressure (mmHg) | 0 [-26 to 10]
  Mean right atrial pressure (mmHg) | 0 [-9 to 6]
  Mean pulmonary capillary wedge pressure (mmHg) | -1.0 [-15 to 8]

2. Secondary Outcome: Change in Exercise Capacity as Measured by the 6-minute Walk Test (6MWT) Over the 24-week Treatment Period.
Description: The 6MWT was conducted at Baseline, 2 to 4 hours after the last Tyvaso dose, and prior to first dose of UT-15C SR. The 6MWT was also performed at Weeks 4, 12, and 24, or at the time of premature termination of study drug if prior to the Week 24 visit.
Time Frame: Baseline and Weeks 4, 12, and 24
Population: Intent-to-treat population with data available at Baseline and Week 24.
Measure: Median (Full Range); unit: Meters
Arm/Group | UT-15C SR BID
Number analyzed (Participants) | 18
Meters
  Week 4 | 20.5 [-111 to 119]
  Week 12 | 12.4 [-70 to 101]
  Week 24: number analyzed (Participants) | 15
  Week 24 | 14.9 [-178 to 101]

3. Secondary Outcome: Time to Clinical Worsening Over the Treatment Period.
Description: Clinical worsening was assessed continuously from Baseline through each subject's last study visit. Clinical worsening was defined as the occurrence of any one or more of the following: death (all causes), hospitalization as a result of worsening pulmonary arterial hypertension (PAH), and initiation of a parenteral prostacyclin.
Time Frame: Clinical worsening was assessed continuously from Baseline through each subject's last study visit
Population: Intent-to-treat population with data available at Baseline and Week 24.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | UT-15C SR BID
Number analyzed (Participants) | 18
Days | 234 (200.3)

4. Secondary Outcome: Shift From Baseline in World Health Organization (WHO) Functional Class Over the 24-week Treatment Period.
Description: The WHO functional classification for pulmonary hypertension was assessed at Baseline prior to starting UT-15C SR, Weeks 4, 8, 12, and 24, or at the time of premature termination if prior to Week 24. The WHO functional classification ranges from I (patient's disease does not affect daily activities) to IV (patient's disease causes severe impairment).
Time Frame: Baseline and Weeks 4, 8, 12, and 24
Population: Intent-to-treat population with data available at Baseline and Week 24.
Measure: Number; unit: participants
Groups:
- Class II to Class II; Class II to Class III; Class III to Class II; Class III to Class III: UT-15C SR BID
Arm/Group | Class II to Class II | Class II to Class III | Class III to Class II | Class III to Class III
Number analyzed (Participants) | 18 | 18 | 18 | 18
participants
  Week 4 | 8 | 1 | 0 | 9
  Week 8 | 6 | 3 | 2 | 7
  Week 12 | 9 | 0 | 1 | 8
  Week 24: number analyzed (Participants) | 15 | 15 | 15 | 15
  Week 24 | 7 | 1 | 2 | 5

5. Secondary Outcome: N-terminal Pro-Brain Natriuretic Peptide (NT-proBNP) Over the 24-week Treatment Period.
Description: NT-proBNP was assessed at Baseline prior to starting UT-15C SR, Weeks 12 and 24, or at the time of premature termination if prior to Week 24. Blood for NT-proBNP assessment was collected before the 6MWT was conducted.
Time Frame: Baseline and Weeks 12 and 24
Population: Intent-to-treat population with data available at Baseline and Week 24.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | UT-15C SR BID
Number analyzed (Participants) | 16
pg/mL
  Week 12 | -99 (295)
  Week 24: number analyzed (Participants) | 13
  Week 24 | 144 (464)

6. Primary Outcome: Change in Hemodynamic Parameter (Heart Rate) From Baseline to Week 24.
Description: Heart rate was assessed at Baseline and Week 24 or at the time of premature termination of study drug if prior to the Week 24 visit.
Time Frame: Baseline and Week 24
Population: Intent-to-treat population with data available at Baseline and Week 24.
Measure: Median (Full Range); unit: beats/min
Arm/Group | UT-15C SR BID
Number analyzed (Participants) | 15
beats/min | 4.00 [-29.0 to 25.0]

7. Primary Outcome: Change in Hemodynamic Parameters (Arterial and Venous Oxygen Saturation) From Baseline to Week 24.
Description: Hemodynamics (via right heart catheterization [RHC]) were assessed at Baseline and Week 24 or at the time of premature termination of study drug if prior to the Week 24 visit.
  Cardiopulmonary hemodynamic measurements included arterial oxygen saturation (SaO2) and mixed venous oxygen saturation (SvO2).
Time Frame: Baseline and Week 24
Population: Intent-to-treat population with data available at Baseline and Week 24.
Measure: Median (Full Range); unit: percentage bound to hemoglobin
Arm/Group | UT-15C SR BID
Number analyzed (Participants) | 15
percentage bound to hemoglobin
  Arterial oxygen saturation (%) | 1.0 [-5 to 5]
  Mixed venous oxygen saturation (%) | 0 [-9 to 4]

8. Primary Outcome: Change in Hemodynamic Parameter (Cardiac Output) From Baseline to Week 24.
Description: Hemodynamics (via right heart catheterization [RHC]) were assessed at Baseline and Week 24 or at the time of premature termination of study drug if prior to the Week 24 visit.
Time Frame: Baseline and Week 24
Population: Intent-to-treat population with data available at Baseline and Week 24.
Measure: Median (Full Range); unit: L/min
Arm/Group | UT-15C SR BID
Number analyzed (Participants) | 15
L/min | 0 [-1 to 4]

9. Primary Outcome: Change in Hemodynamic Parameter (Cardiac Index) From Baseline to Week 24.
Description: Hemodynamics (via right heart catheterization [RHC]) were assessed at Baseline and Week 24 or at the time of premature termination of study drug if prior to the Week 24 visit.
  Cardiopulmonary hemodynamic measurements included cardiac index (CI).
Time Frame: Baseline and Week 24
Population: Intent-to-treat population with data available at Baseline and Week 24.
Measure: Median (Full Range); unit: L/min/m^2
Arm/Group | UT-15C SR BID
Number analyzed (Participants) | 15
L/min/m^2 | 0 [0 to 1]

10. Primary Outcome: Change in Hemodynamic Parameter (Pulmonary Vascular Resistance Index) From Baseline to Week 24.
Description: Hemodynamics (via right heart catheterization [RHC]) were assessed at Baseline and Week 24 or at the time of premature termination of study drug if prior to the Week 24 visit.
  Cardiopulmonary hemodynamic measurements included the following: pulmonary vascular resistance index (PVRI).
Time Frame: Baseline and Week 24
Population: Intent-to-treat population with data available at Baseline and Week 24.
Measure: Median (Full Range); unit: dyn*s/cm^5*m^2
Arm/Group | UT-15C SR BID
Number analyzed (Participants) | 15
dyn*s/cm^5*m^2 | 0.2 [-10 to 7]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded throughout the 24-week study, including the screening phase, as well as during the long-term follow-up period.
Description: Adverse events were recorded throughout the course of the study, including a 24-week treatment period and a long-term follow up period through each subject's last study visit (up to 553 days).
Arm/Group | UT-15C SR BID
Serious Adverse Events (participants affected / at risk) | 2/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UT-15C SR BID (N=18)
Ascites (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UT-15C SR BID (N=18)
Diarrhea (Gastrointestinal disorders) | 11 (11)
Headache (Nervous system disorders) | 14 (14)
Nausea (Gastrointestinal disorders) | 12 (12)
Flushing (Vascular disorders) | 8 (8)
Fatigue (General disorders) | 6 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Edema peripheral (General disorders) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Chest discomfort (General disorders) | 3 (3)
Chest pain (General disorders) | 3 (3)
Hypotension (Vascular disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasopharyngitis (Infections and infestations) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Blood urea increased (Investigations) | 2 (2)
Bronchitis (Infections and infestations) | 2 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2)
Presyncope (Nervous system disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Sinusitis (Infections and infestations) | 2 (3)
Syncope (Nervous system disorders) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (3)
Anxiety (Psychiatric disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Atrial fibrillatioin (Cardiac disorders) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Chills (General disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Duodenal polyp (Gastrointestinal disorders) | 1 (1)
Dysguesia (Nervous system disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eye burns (Injury, poisoning and procedural complications) | 1 (1)
Face edema (General disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hematocrit decreased (Investigations) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hemoglobin decreased (Investigations) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Local swelling (General disorders) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Edema (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Red blood cell count decreased (Investigations) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Weight increased (Investigations) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Affect lability (Psychiatric disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator agree not to publish or publicly present any interim results of the study without the prior written consent of Sponsor, not to be unreasonably withheld or delayed, except as provided below. Institution and/or Principal Investigator further agree to provide Sponsor with drafts of any such publication or presentation for review and approval no less than 30 days prior to submission for publication or the date of public presentation.